CLINICAL TRIAL: NCT05191147
Title: Prevalence of Dietary Supplement Consumption Among Pregnant Women During the First 20-25 Weeks of Pregnancy: a Cross-sectional Telephone Interview Survey
Brief Title: Prevalence of Dietary Supplement Consumption Among Pregnant Womenweeks of Pregnancy: a Cross-sectional Telephone Interview Survey
Acronym: PCAFE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.0368
Record Dates: First submitted 2021-12-22; First posted 2022-01-13 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Preference, Consumer
MeSH Terms: conditions — Consumer Behavior | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Dietary supplement — We will study dietary supplement consumption among pregnant women

SUMMARY:
Primary endpoint :

Prevalence estimation of the dietary supplement consumption among pregnant women during the first 20-25 weeks of pregnancy.

Hypothesis of the study :

The sale and consumption of dietary supplements in the general population has increased in recent years. It would be interesting to know if this is also the case for pregnant women or if they are more vigilant about their health during this period. It would also allow to identify factors associated with their consumption if it exists.

The investigators hypothesize that some women may sometimes fail to mention this supplement intake to care givers and they would like to know if these omissions are voluntary or not.

DETAILED DESCRIPTION:
Dietary supplement are foodstuffs whose purpose is to supplement the normal diet, by constituting a concentrated source of nutrients or other substances with a nutritional or physiological effect, alone or in combination. There are many dietary supplement, based on plants, vitamins and minerals, or other concentrates of substances with a nutritional and physiological purpose.

Thus, the consumption of dietary supplement in pregnant women is interesting to pursue because no prevalence exists on the general consumption of food supplements in pregnant women in early pregnancy. Only studies on diet and the potential danger of supplements have been carried out. More specific studies on certain types of vitamins have also been carried out but no prevalence on general consumption has been found.

Therefore, the aim of the study is to know the extent of dietary supplementation in early pregnancy, and the associated factors in order to take it into account in the management and follow-up of patients. The investigators would also like to know the intentions and motivations of these women to consume these products.

To proceed, they will give an information sheet that will allow the collection of the telephone number, during an ultrasound (between 20 and 25 weeks of amenorrhea).Then they will call them and during the telephone interview, they will collect informations needed.

Distribution of an information sheet that will allow the collection of the telephone number of each patient coming for their second trimester ultrasound (between 20 and 25 SA). This form will be accompanied by the letter of information and non-objection which will be kept by the patient. The distribution will be done by the health professionals performing the ultrasound at the beginning or at the end of the medical appointment.

So, the primary endpoint is the proportion of women who report taking at least one dietary supplement during the first 20-25 weeks of pregnancy. This information will be collected by a phone interview.

The secondary endpoints are :

* Describe the dietary supplements consumed during the first 20-25 weeks of pregnancy: galenic form, indication, source of information, place of purchase (pharmacy, supermarket etc.)
* Assess whether beliefs about medication are associated with the use of dietary supplements during pregnancy, using BMQ (Belief on Medicine Questionnaire)
* Describe the mean number of dietary supplements taken by patients in early pregnancy
* Describe the frequency of use for each dietary supplement ('(several times a day / once a day /several times a week / once a week / once a month etc...)

ELIGIBILITY:
Inclusion Criteria:

* Aged of 18 or older
* Pregnant woman
* Performing a 2nd trimester ultrasound between 20 and 25 ammenorhea week
* Informed consent signed
* Affiliated to social security insurance or beneficiary of social security insurance

Exclusion Criteria:

* Subject participating in another study
* Subject under administrative or legal supervision
* Non-speaking french
* Opposing their participation in the research

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant woman who come in the service for an ultrasound
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-10 (Estimated); Study Completion 2022-05-10 (Estimated)

PRIMARY OUTCOMES:
the proportion of women who report taking at least one dietary supplement during the first 20-25 weeks of pregnancy | 1 month
  what is the percentage of pregnant women who take dietary supplement

SECONDARY OUTCOMES:
Describe the dietary supplements consumed during the first 20-25 weeks of pregnancy | 1 month
  Which galenic form, indication, source of information, place of purchase (pharmacy, supermarket etc.)
Assess whether beliefs about medication are associated with the use of dietary supplements during pregnancy | 1 month
  using BMQ (Belief on Medicine Questionnaire)
Describe the mean number of dietary supplements taken by patients in early pregnancy | 1 month
  How many dietary supplement pregnant women take on a daily basis
Describe the frequency of use for each dietary supplement | 1 month
  Several times a day / once a day /several times a week / once a week / once a month etc.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No